CLINICAL TRIAL: NCT06699966
Title: Stony Brook Medicine Anti-Inflammatory Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Ramin Parsey, Principle Investigator (M.D., Ph.D.), Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00259
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Celecoxib; Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Celecoxib Arm (Experimental): Participants will take 400mg (two 200mg tablets) of celecoxib daily with a meal for 8 weeks.
  Interventions: Drug: Celecoxib
- Minocycline (Experimental): Participants will take minocyline for 8 weeks. Dosing of minocycline will gradually increase from 50 mg per day during Week 1, increase to 50 mg b.i.d. during Week 2, and finally reach 100 mg b.i.d. during Weeks 3-8.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Celecoxib — The dose of celecoxib will be at the maximum recommended FDA approved dose (400mg daily). Participants will take two 200mg tablets of celecoxib daily with a meal for 8 weeks.
  Other Names: Celebrex
  Arms: Celecoxib Arm
Drug: Minocycline — Dosing of minocycline will gradually increase from 50 mg per day during Week 1, increase to 50 mg b.i.d. during Week 2, and finally reach 100 mg b.i.d. during Weeks 3-8.
  Arms: Minocycline

SUMMARY:
This is an experimental study designed to measure the effect of celecoxib or minocycline on depressive symptoms in unipolar and bipolar depression. Participants will be equally randomized to either celecoxib or minocycline. All participants will complete a battery of clinical and psychological assessments prior to treatment assignment, and again after treatment completion, to assess any changes or improvements in depression.

ELIGIBILITY:
Inclusion Criteria:

* Current consent form signed
* Capacity to give informed consent
* Age range 18-65 (inclusive)
* Diagnosis of MDD or bipolar depression and currently in a major depressive episode
* Score of at least 29 on the MADRS (at least moderate depression)

Exclusion Criteria:

* Hypersensitivity to celecoxib, minocycline, tetracyclines, sulfonamides, aspirin, other NSAIDs, or any component of the formulation; previous asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs
* History of myocardial infarction or current cardiac condition
* Heptic impairment, heart failure, severe renal impairment, recent GI bleed, history of peptic ulcer disease, anemia or any other contraindication for celecoxib or minocycline
* Poor CYP2C9 metabolizer
* Currently taking medications that interact with celecoxib (digoxin, antihypertensives, diuretics, anticoagulant or anti-platelet treatment, including aspirin), or minocycline (isotretinoin, ergot alkaloids) without providing physicians approval
* Use of herbs, drugs, or medications with anti-inflammatory or immunomodulatory properties (within 5 half-lives of starting celecoxib or minocycline treatment)
* Unlikely to tolerate medication washout or the medication-free period following washout.
* Participant considered at significant risk for suicide.
* Electroconvulsive therapy (ECT) within 1 month
* High potential for excessive drug/alcohol use during the treatment period (excluding nicotine or cannabis)
* Significant active physical illness or neurological deficit that may affect brain functioning.
* If participant is currently pregnant, breastfeeding, or planning to conceive during the course of study participation.
* Need for medications that control mania.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Hamilton Depression Rating Scale (HAM-D 24) Score at 8 Weeks | Baseline and 8 weeks.
  Participants will have a Hamilton Depression Rating Scale-24 (HDRS) score obtained at baseline. Minimum score 0, maximum possible score 75; the higher the score on the scale, the more severe the degree of depression. After eight weeks of medication treatment, the HDRS score will be reevaluated with the HDRS-24. Participants who have a 50% or greater decrease in their HDRS-24 score will be considered responders (to treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Parsey, M.D, Ph.D., Principal Investigator — Stony Brook University